CLINICAL TRIAL: NCT06134817
Title: Prospective Pilot Study on Geniculate Artery Embolization for Treatment of Persistent Knee Pain Post Total Knee Arthroplasty
Brief Title: Geniculate Artery Embolization for Treatment of Persistent Knee Pain Post Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of PI.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-00595
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Knee Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients with Post TKA Knee Pain (Experimental): Patients with persistent knee pain resistant to conservative management for at least 9 months after total knee arthroplasty (TKA) will receive geniculate artery embolization (GAE) using Embozene Color-Advanced Microspheres. Treatment will be completed during one interventional session.
  Interventions: Device: Embozene Color-Advanced Microspheres.

INTERVENTIONS:
Device: Embozene Color-Advanced Microspheres. — Embozene Microspheres are spherical, tightly calibrated, biocompatible, nonresorbable, hydrogel microspheres coated with an inorganic perfluorinated polymer. The microspheres are intended to occlude vasculature for the purpose of blocking blood flow to a target tissue.
  In the study, the abnormal vessels will be embolized with 100 μm Embozene Microspheres solution under direct fluoroscopic visualization to prevent reflux and non-target embolization. Multiple geniculate arteries may be embolized until neovascularity is no longer seen.

SUMMARY:
Single-arm, single-center, no sham or placebo, prospective pilot trial designed to evaluate the safety and efficacy of transcatheter arterial embolization in patients with persistent knee pain resistant to conservative management for at least 9 months after total knee arthroplasty (TKA). Eligible participants will receive geniculate artery embolization (GAE) using Embozene™ Color-Advanced Microspheres. Patients will be followed up for a total of 24 months after GAE.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain resistant to conservative treatment for at least 9 months post TKA performed for knee OA, and
* Moderate to severe knee pain: pain VAS ≥40 mm, and
* Willing, able, and mentally competent to provide informed consent and complete study questionnaires in English. The Study questionnaires are validated in English.

Exclusion Criteria:

* Active systemic or local knee infection or;
* Active malignancy or;
* Life expectancy less than 6 months or;
* Prior ipsilateral knee arthroscopic surgery or repeat TKA (within 9 months of screening) or;
* Ipsilateral knee intra-articular injection in the last 3 months or;
* Rheumatoid arthritis, spondyloarthropathies, crystal disease, gout, pseudogout, or lupus or;
* Pregnant during the study period or;
* Renal dysfunction as defined by serum creatinine >1.6 dl/mg or eGFR <60 on blood tests obtained within 30 days of procedure or;
* Body weight greater than 200 Kg or;
* Known history of severe contrast allergy to iodinated contrast resulting in anaphylaxis or;
* Known significant arterial atherosclerosis that would limit selective angiography and/or lower extremity symptoms thought to be secondary to arterial vascular disease (eg claudication, ischemic rest pain) or;
* known avascular necrosis in the target knee or;
* Complications of TKA such as suspected or confirmed early loosening, ligamentous instability, reflex sympathetic dystrophy, polyethylene wear with or without particle disease (osteolysis), and large effusions (with or without hemarthrosis) or;
* Patient is enrolled in a different trial for treatment of knee pain post total knee arthroplasty (ipsilateral knee)

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bedros Taslakian, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Bedros.Taslakian@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Bedros.Taslakian@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note that while the Protocol Enrollment is N=2, N=1 participant was a screen failure and did not begin the study. Thus, the Number of Participants started is N=1.
Groups:
- Patients With Post TKA Knee Pain: Patients with persistent knee pain resistant to conservative management for at least 9 months after total knee arthroplasty (TKA) will receive geniculate artery embolization (GAE) using Embozene Color-Advanced Microspheres. Treatment will be completed during one interventional session.
  Embozene Color-Advanced Microspheres.: Embozene Microspheres are spherical, tightly calibrated, biocompatible, nonresorbable, hydrogel microspheres coated with an inorganic perfluorinated polymer. The microspheres are intended to occlude vasculature for the purpose of blocking blood flow to a target tissue.
  In the study, the abnormal vessels will be embolized with 100 μm Embozene Microspheres solution under direct fluoroscopic visualization to prevent reflux and non-target embolization. Multiple geniculate arteries may be embolized until neovascularity is no longer seen.
Period: Overall Study
Arm/Group | Patients With Post TKA Knee Pain
Started | 1
Completed | 0
Not Completed | 1
Not completed — Physician Departure - termination of study | 1

BASELINE CHARACTERISTICS:
Population: N= 1 participant was a screen failure; thus, baseline characteristics are presented for the N= 1 participant who entered the study and was treated.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (NA) — N=1 participant.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Score From Baseline to Month 6
Description: The Pain subscale of the KOOS consists of 9 items measuring pain associated with the knee. Each item is rated on a Likert scale from 0 (No Problems) to 4 (Extreme Problems). The raw score is the sum of responses and is transformed to a 0-100 scale, where zero represents extreme knee problems and 100 represents no knee problems.
Time Frame: Baseline, Month 6 Post-GAE Procedure
Measure: Number; unit: Percent change in KOOS Pain score
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 1
Percent change in KOOS Pain score | 20

2. Secondary Outcome: Change From Baseline in KOOS Symptoms Score
Description: The Symptoms subscale of the KOOS consists of 7 items measuring symptoms associated with the knee. Each item is rated on a Likert scale from 0 (No Problems) to 4 (Extreme Problems). The raw score is the sum of responses and is transformed to a 0-100 scale, where zero represents extreme knee problems and 100 represents no knee problems.
Time Frame: Baseline, Month 3 Post-GAE Procedure
Measure: Number; unit: Percentage change in KOOS Symptoms score
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 1
Percentage change in KOOS Symptoms score | 23

3. Secondary Outcome: Change From Baseline in KOOS Symptoms Score
Description: as for outcome 2
Time Frame: Baseline, Month 6 Post-GAE Procedure
Measure: Number; unit: Percentage change in KOOS Symptoms score
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 1
Percentage change in KOOS Symptoms score | 31

4. Secondary Outcome: Change From Baseline in KOOS Symptoms Score
Description: as for outcome 2
Time Frame: Baseline, Month 12 Post-GAE Procedure
Population: Patient did not complete necessary follow-up visit to collect measure data.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in KOOS Symptoms Score
Description: as for outcome 2
Time Frame: Baseline, Month 24 Post-GAE Procedure
Population: Patient did not complete necessary follow-up visit to collect measure data.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Knee Pain Measured Via Visual Analogue Scale (VAS)
Description: The VAS measures knee pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). The patient uses a ruler to measure the distance in centimeters from the 'no pain marker' (or zero) to the current pain mark. This provides a pain intensity score out of 10; for example, 6 out of 10 (or 6/10). Higher scores indicate greater knee pain.
Time Frame: Baseline, Month 3 Post-GAE Procedure
Measure: Number; unit: Percentage change in VAS score
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 1
Percentage change in VAS score | 42

7. Secondary Outcome: Change From Baseline in Knee Pain Measured Via VAS
Description: as for outcome 6
Time Frame: Baseline, Month 6 Post-GAE Procedure
Measure: Number; unit: Percentage change in VAS score
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 1
Percentage change in VAS score | 46

8. Secondary Outcome: Change From Baseline in Knee Pain Measured Via VAS
Description: as for outcome 6
Time Frame: Baseline, Month 12 Post-GAE Procedure
Population: Patient did not complete necessary follow-up visit to collect measure data.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline in Knee Pain Measured Via VAS
Description: as for outcome 6
Time Frame: Baseline, Month 24 Post-GAE Procedure
Population: Patient did not complete necessary follow-up visit to collect measure data.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in Quality of Life Measured Via EuroQol-5 Dimension-5 Level (EQ-5D-5L) Score
Description: Patient Reported Outcome (PRO) instrument that uses 6 questions to generally assess patients' quality of life. The EQ-5D-5L system defines so-called EQ5D Health States; depending on the level, a number is assigned to each dimension, so that a 5-digit number combination is obtained. This 5-digit number is converted into a score using an algorithm. This point value is called the EQ-5D-5L index. An index value of 1 represents the best possible quality of life, while an index value of <0 represents the worst possible quality of life.
Time Frame: Baseline, Month 3 Post-GAE Procedure
Population: Outcome data not collected at Month 3 timepoint.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline in Quality of Life Measured Via EQ-5D-5L Score
Description: as for outcome 10
Time Frame: Baseline, Month 6 Post-GAE Procedure
Measure: Number; unit: Percentage change in EQ-5D-5L score
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 1
Percentage change in EQ-5D-5L score | 19

12. Secondary Outcome: Change From Baseline in Quality of Life Measured Via EQ-5D-5L Score
Description: as for outcome 10
Time Frame: Baseline, Month 12 Post-GAE Procedure
Population: Patient did not complete necessary follow-up visit to collect measure data.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 0

13. Secondary Outcome: Change From Baseline in Quality of Life Measured Via EQ-5D-5L Score
Description: as for outcome 10
Time Frame: Baseline, Month 24 Post-GAE Procedure
Population: Patient did not complete necessary follow-up visit to collect measure data.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 0

14. Secondary Outcome: Incidence of Synovitis
Description: Incidence of synovitis measured using magnetic resonance angiogram images.
Time Frame: Month 6 Post-GAE Procedure
Population: Outcome not assessed.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 0

15. Secondary Outcome: Incidence of Synovitis
Description: Incidence of synovitis measured using magnetic resonance angiogram images.
Time Frame: Month 24 Post-GAE Procedure
Population: Patient did not complete necessary follow-up visit to collect measure data.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 0

16. Secondary Outcome: Incidence of Successful Selective Catheterization of Target Genicular Artery
Time Frame: Up to Month 24 Post-GAE Procedure
Population: Patient did not complete necessary follow-up visit to collect measure data.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 0

17. Secondary Outcome: Incidence of Successful Embolization From at Least One Feeding Artery of the Knee Joint
Description: Successful embolization defined as suppression or reduction in the filling of (blood flow in) abnormal vessels visible on angiography.
Time Frame: Up to Month 24 Post-GAE Procedure
Population: Patient did not complete necessary follow-up visit to collect measure data.
Arm/Group | Patients With Post TKA Knee Pain
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months.
Description: The PI recorded all reportable events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. At each study visit, the investigator inquired about the occurrence of AE/SAEs since the last visit. Events were followed for outcome information until resolution or stabilization.
Arm/Group | Patients With Post TKA Knee Pain
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT06134817/Prot_SAP_000.pdf